CLINICAL TRIAL: NCT04465149
Title: Comparative Study of the Anaesthetic Efficacy of 4% Articaine Versus 2% Mepivacaine in Mandibular Third Molar Germectomy Using Different Anaesthetic Techniques: a Split-mouth Clinical Trial
Brief Title: Efficacy of Differents Anaesthetics in Mandibular Third Molar Germectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alfredo De Rosa, Associated Professor, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SecondUNI-1
Record Dates: First submitted 2020-05-07; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Local Anesthetic Efficacy

STUDY DESIGN:
Intervention Model Description: The subjects were children undergoing orthodontic treatment in whom early extraction was indicated to facilitate their treatment in some specific conditions (i.e. posterior crowding, altered second molar eruption, non-extraction approach). For each subject, the first germectomy was scheduled 15 days apart. The same senior operator, assisted by the same practitioner, completed all the surgical procedures. All interventions made with mepivacaine were performed with the same anaesthetic technique routinely used in Oral surgery (IANB). The technique was complemented with anaesthesia of the buccal nerve, as routine for this technique, administering another 1.8 ml of the same anaesthetic used in each intervention. On the other hand, the surgical procedures in articaine cases were made practising a plexus technique, performing a deep buccal injection distally to the second mandibular molar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients who required germectomy of mandibular third molars. Each patient received local anaesthesia on one side with articaine inoculated with plexus technique while on the other side with mepivacaine using inferior alveolar nerve block technique.
  Interventions: Procedure: Third Molar Germectomy

INTERVENTIONS:
Procedure: Third Molar Germectomy — Surgical extraction of Third Molars that exhibits at least a third of its root in formation, with a periodontal ligament discernible on panoramic x-ray (defined as germectomy).

SUMMARY:
Aim: To compare the clinical efficacy of local anaesthetics with articaine 4% or mepivacaine 2% (both with epinephrine 1:100.000) using different anaesthetic techniques to perform germectomy of lower third molars and to assess patients' feelings and pain during surgery.

Methods: 50 patients (ranged 11-16 years) who required germectomy of mandibular third molars were recruited. Each patient received local anaesthesia on one side with articaine inoculated with plexus technique while on the other side with mepivacaine using inferior alveolar nerve block technique. The patients' evaluation was performed on pre and intraoperative tactile-pressure feelings and intraoperative pain with four levels on the analogic visual scale (VAS).

DETAILED DESCRIPTION:
The surgical extraction of a tooth that exhibits at least a third of its root in formation, with a periodontal ligament discernible on panoramic x-ray, is defined as germectomy. Early germectomy is a usefull intervention to avoid problems caused by lower third molar retention and impaction, and it is often required before or after orthodontic treatment. This surgical technique would also allow to avoid complications, such as inferior alveolar and lingual nerve damage.

The control of the patient's pain and anxiety by using local anaesthesia is essential in oral surgery: these aspects become more important in adolescents, above all in the case of third molar germectomy. Local anaesthetic (LA) injection is often the only painfull part of the dental procedure, and the fear associated with this technique is the main reason that leads patients to avoid dental treatment.

During the execution of dental surgical procedures, anaesthesia of the structures innervated by the mandibular nerve is necessary, and many local anaesthetic techniques are described in the literature. Generally, infiltration plexus technique is usually performed for maxillary procedures while IANB is used for molar mandibular sites with 2% local anaesthetics. Failure rates for IANB are high, sometimes reaching 80% for the lower incisors with this technique, and numerous approaches for the implementation of a new technique of IANB have been described. Among them, the articaine 4% already has been successfully used to achieve local anesthesia and facial infiltration anaesthetic technique in the mandible showed efficacy with encouraging result that can be overlapped to the IANB technique. Articaine (4-methyl-3-[2-(propylamino)-propionamido]-2-thiophene-carboxylic acid, methyl ester hydrochloride) contains a thiophene ring instead of benzene and an ester group. The thiophene ring allows for higher lipid solubility so a greater portion of an administered dose can enter in neurons. Gazal found that a combination of nerve block anaesthesia, buccal infiltration and intra-ligamentary injection resulted in more profound anaesthesia (P =0.003) and higher success rates compared to IANB alone in mandibular first molar pulp anaesthesia. Other studies reported the use of articaine in implantology interventions in which it was used with subperiosteal technique on the buccal and vestibular sides.

Thus, the literature showed several conflicting results on the mandibular facial plexus infiltration technique used with different anesthetics.

Recent studies of this anaesthetic technique found that 1.8 cc of 4% articaine facial infiltration in the mandible can be effective when the thickness of mandibular facial cortex is < 2.0-3.0 mm, with 5-10 minutes needed for the adequate anaesthesia.

It was reported that many dental procedures on deciduous molars could be accomplished with infiltration of articaine alone in the pediatric population.

As above mentioned, the difficulty in achieving reliable anaesthesia in the third mandibular molars in adults with facial infiltration of local anaesthetic is related to the thickness of the cortical bone and inability to achieve consistently inferior alveolar nerve.

An ideal local anaesthetic should have the following characteristics:

1. short latency time;
2. strength of the intense effect;
3. duration of prolonged action;
4. lack of harmful local and systemic effects. Currently, mepivacaine is among the most used and studied anaesthetics in dentistry; however, articaine is nowadays increasingly used for its manageability, lack of side effects and high anaesthetic potency. Mepivacaine is an amide-type anaesthetic with fast action from the beginning and 30-120 minutes duration. Its maximum allowed dose is 300 mg with epinephrine or 500 mg alone. The dose for children is 4-6 mg/kg/dose (maximum: 270 mg) without epinephrine.

Articaine, due to its chemical characteristics, is quickly soluble and rapidly released from adipose/lipid tissue. The ester side chain of articaine is hydrolyzed by plasmaesterases rendering the molecule inactive. Evidence suggests that it is the local anaesthetic that best spreads within soft and hard tissues. Then, it has a non-conducive effect on extended operations having a shorter half-life of 25 minutes compared to approximately 90 minutes of other amides (115 minutes for mepivacaine) that require hepatic clearance. Accordingly, it was suggested that articaine does not own any relevant side effects or systemic toxicities.

For this reason, articaine has been used at higher concentrations (4%), associated with epinephrine, compared to other local dental anesthetics. This higher concentration ensures an excellent spread both in hard and soft tissues, also promoted by a pKa very similar to the physiological pH of tissues. Its great liposolubility allows a rapid diffusion in adipose tissue (spread coefficient = 17,0) and involves a lower adherence to the nerve membranes and, above all, lower toxicity for the tissues. Moreover, articaine has a high protein-based bond (94%) which allows a better affinity for the protein-based membrane receptors, and it is a direct sign of its increased anaesthetic potency.

Dental local anaesthetics are often combined with vasoconstrictors, such as epinephrine, to increase the depth and duration of analgesia. Clinical experiments, in which articaine without vasoconstrictor was used, did not show any satisfying results, whereas the use of articaine combined with low concentrations of vasoconstrictors produced better anaesthetic effects than other common local anaesthetics such as bupivacaine and mepivacaine. It is well documented that vasoconstrictors have a safety range if used at low doses, and not directly injected in the blood vessels, even in particular care patients.

The present study aimed to compare the clinical efficacy of articaine 4% (epinephrine 1:100.000) versus mepivacaine 2% (epinephrine 1:100.000) for the surgical germectomy of mandibular third molars with two different conventional anaesthetic techniques in young patients whom jawbone is not completely mineralized yet and more penetrable by the articaine molecule.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring bilateral germectomy of mandibular third molars before orthodontic treatment

Exclusion Criteria:

* Patients presenting systemic and oral diseases

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
Discomfort/Pain felt for anesthetic injection valued by the Patient on a Visual Analogue Scale | At the beginning of Surgery
  Once performed the injections, patients were asked to notice on a visual analogue scale, how much discomfort they felt due to the anaesthetic injections, indicating one of the following values:
  0 absent
  1. mild
  2. moderate
  3. severe

SECONDARY OUTCOMES:
Test during the Surgery | After 10/15 minutes
  The same test was repeated intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Marco Menditti, Doctor, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania Luigi Vanvitelli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perillo L, Vitale M, d'Apuzzo F, Isola G, Nucera R, Matarese G. Interdisciplinary approach for a patient with unilateral cleft lip and palate. Am J Orthod Dentofacial Orthop. 2018 Jun;153(6):883-894. doi: 10.1016/j.ajodo.2016.12.035. PMID 29853246
- [Result] Raucci G, Pacheco-Pereira C, Elyasi M, d'Apuzzo F, Flores-Mir C, Perillo L. Short- and long-term evaluation of mandibular dental arch dimensional changes in patients treated with a lip bumper during mixed dentition followed by fixed appliances. Angle Orthod. 2016 Sep;86(5):753-60. doi: 10.2319/073015-519.1. Epub 2016 Jan 15. PMID 26771718
- [Result] Chiapasco M, Crescentini M, Romanoni G. [The extraction of the lower third molars: germectomy or late avulsion?]. Minerva Stomatol. 1994 May;43(5):191-8. Italian. PMID 8072466
- [Result] Rayati F, Noruziha A, Jabbarian R. Efficacy of buccal infiltration anaesthesia with articaine for extraction of mandibular molars: a clinical trial. Br J Oral Maxillofac Surg. 2018 Sep;56(7):607-610. doi: 10.1016/j.bjoms.2018.06.012. Epub 2018 Jul 3. PMID 29980352
- [Result] Almpani K, Kolokitha OE. Role of third molars in orthodontics. World J Clin Cases. 2015 Feb 16;3(2):132-40. doi: 10.12998/wjcc.v3.i2.132. PMID 25685759
- [Result] Bjornland T, Haanaes HR, Lind PO, Zachrisson B. Removal of third molar germs. Study of complications. Int J Oral Maxillofac Surg. 1987 Aug;16(4):385-90. doi: 10.1016/s0901-5027(87)80072-3. PMID 3117908
- [Result] Eccleston C. Role of psychology in pain management. Br J Anaesth. 2001 Jul;87(1):144-52. doi: 10.1093/bja/87.1.144. PMID 11460803
- [Result] Gunter JB. Benefit and risks of local anesthetics in infants and children. Paediatr Drugs. 2002;4(10):649-72. doi: 10.2165/00128072-200204100-00003. PMID 12269841
- [Result] Milgrom P, Coldwell SE, Getz T, Weinstein P, Ramsay DS. Four dimensions of fear of dental injections. J Am Dent Assoc. 1997 Jun;128(6):756-66. doi: 10.14219/jada.archive.1997.0301. PMID 9188235
- [Result] Kaufman E, Epstein JB, Naveh E, Gorsky M, Gross A, Cohen G. A survey of pain, pressure, and discomfort induced by commonly used oral local anesthesia injections. Anesth Prog. 2005 Winter;52(4):122-7. doi: 10.2344/0003-3006(2005)52[122:ASP]2.0.CO;2. PMID 16596910
- [Result] Khoury J, Townsend G. Neural blockade anaesthesia of the mandibular nerve and its terminal branches: rationale for different anaesthetic techniques including their advantages and disadvantages. Anesthesiol Res Pract. 2011;2011:307423. doi: 10.1155/2011/307423. Epub 2011 May 25. PMID 21716730
- [Result] Flanagan DF. The effectiveness of articaine in mandibular facial infiltrations. Local Reg Anesth. 2015 Dec 18;9:1-6. doi: 10.2147/LRA.S94647. eCollection 2016. PMID 26730209
- [Result] Saxena P, Gupta SK, Newaskar V, Chandra A. Advances in dental local anesthesia techniques and devices: An update. Natl J Maxillofac Surg. 2013 Jan;4(1):19-24. doi: 10.4103/0975-5950.117873. PMID 24163548
- [Result] Meechan JG. The use of the mandibular infiltration anesthetic technique in adults. J Am Dent Assoc. 2011 Sep;142 Suppl 3:19S-24S. doi: 10.14219/jada.archive.2011.0343. PMID 21881058
- [Result] Malamed SF. Is the mandibular nerve block passe? J Am Dent Assoc. 2011 Sep;142 Suppl 3:3S-7S. doi: 10.14219/jada.archive.2011.0340. PMID 21881055
- [Result] Gazal G, Fareed WM, Zafar MS. Role of intraseptal anesthesia for pain-free dental treatment. Saudi J Anaesth. 2016 Jan-Mar;10(1):81-6. doi: 10.4103/1658-354X.169482. PMID 26955316
- [Result] Heller AA, Shankland WE 2nd. Alternative to the inferior alveolar nerve block anesthesia when placing mandibular dental implants posterior to the mental foramen. J Oral Implantol. 2001;27(3):127-33. doi: 10.1563/1548-1336(2001)0272.3.CO;2. PMID 12500871
- [Result] Leith R, Lynch K, O'Connell AC. Articaine use in children: a review. Eur Arch Paediatr Dent. 2012 Dec;13(6):293-6. doi: 10.1007/BF03320829. PMID 23235128
- [Result] Gazal G. Comparison of speed of action and injection discomfort of 4% articaine and 2% mepivacaine for pulpal anesthesia in mandibular teeth: A randomized, double-blind cross-over trial. Eur J Dent. 2015 Apr-Jun;9(2):201-206. doi: 10.4103/1305-7456.156811. PMID 26038650
- [Result] Cowan A. Clinical assessment of a new local anesthetic agent-carticaine. Oral Surg Oral Med Oral Pathol. 1977 Feb;43(2):174-80. doi: 10.1016/0030-4220(77)90153-0. PMID 264643
- [Result] Srisurang S, Narit L, Prisana P. Clinical efficacy of lidocaine, mepivacaine, and articaine for local infiltration. J Investig Clin Dent. 2011 Feb;2(1):23-8. doi: 10.1111/j.2041-1626.2010.00035.x. Epub 2010 Nov 8. PMID 25427324
- [Result] Vree TB, Gielen MJ. Clinical pharmacology and the use of articaine for local and regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):293-308. doi: 10.1016/j.bpa.2004.12.006. PMID 15966499
- [Result] Jastak JT, Yagiela JA. Vasoconstrictors and local anesthesia: a review and rationale for use. J Am Dent Assoc. 1983 Oct;107(4):623-30. doi: 10.14219/jada.archive.1983.0307. No abstract available. PMID 6355236
- [Result] Leuschner J, Leblanc D. Studies on the toxicological profile of the local anaesthetic articaine. Arzneimittelforschung. 1999 Feb;49(2):126-32. doi: 10.1055/s-0031-1300372. PMID 10083981
- [Result] Abazarpoor R, Parirokh M, Nakhaee N, Abbott PV. A Comparison of Different Volumes of Articaine for Inferior Alveolar Nerve Block for Molar Teeth with Symptomatic Irreversible Pulpitis. J Endod. 2015 Sep;41(9):1408-11. doi: 10.1016/j.joen.2015.05.015. Epub 2015 Jul 3. PMID 26149210
- [Result] Mittal M, Sharma S, Kumar A, Chopra R, Srivastava D. Comparison of Anesthetic Efficacy of Articaine and Lidocaine During Primary Maxillary Molar Extractions in Children. Pediatr Dent. 2015 Nov-Dec;37(7):520-4. PMID 26883609
- [Result] Corbett IP, Kanaa MD, Whitworth JM, Meechan JG. Articaine infiltration for anesthesia of mandibular first molars. J Endod. 2008 May;34(5):514-8. doi: 10.1016/j.joen.2008.02.042. PMID 18436027
- [Result] Pellicer-Chover H, Cervera-Ballester J, Sanchis-Bielsa JM, Penarrocha-Diago MA, Penarrocha-Diago M, Garcia-Mira B. Comparative split-mouth study of the anesthetic efficacy of 4% articaine versus 0.5% bupivacaine in impacted mandibular third molar extraction. J Clin Exp Dent. 2013 Apr 1;5(2):e66-71. doi: 10.4317/jced.50869. eCollection 2013 Apr 1. PMID 24455059
- [Result] Ram D, Peretz B. Administering local anaesthesia to paediatric dental patients -- current status and prospects for the future. Int J Paediatr Dent. 2002 Mar;12(2):80-9. doi: 10.1046/j.1365-263x.2002.00343.x. PMID 11966886
- [Result] Becker DE, Reed KL. Local anesthetics: review of pharmacological considerations. Anesth Prog. 2012 Summer;59(2):90-101; quiz 102-3. doi: 10.2344/0003-3006-59.2.90. PMID 22822998
- [Result] Vigen EC, Lasse A. Articaine hydrochloride: is it the solution? Dent Update. 2015 Jun;42(5):493. doi: 10.12968/denu.2015.42.5.493. No abstract available. PMID 26964452
- [Result] Kammerer PW, Palarie V, Daublander M, Bicer C, Shabazfar N, Brullmann D, Al-Nawas B. Comparison of 4% articaine with epinephrine (1:100,000) and without epinephrine in inferior alveolar block for tooth extraction: double-blind randomized clinical trial of anesthetic efficacy. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Apr;113(4):495-9. doi: 10.1016/j.tripleo.2011.04.037. Epub 2011 Aug 6. PMID 22676931
- [Result] Pabst L, Nusstein J, Drum M, Reader A, Beck M. The efficacy of a repeated buccal infiltration of articaine in prolonging duration of pulpal anesthesia in the mandibular first molar. Anesth Prog. 2009 Winter;56(4):128-34. doi: 10.2344/0003-3006-56.4.128. PMID 20020793
- [Result] Dudkiewicz A, Schwartz S, Laliberte R. Effectiveness of mandibular infiltration in children using the local anesthetic Ultracaine (articaine hydrochloride). J Can Dent Assoc. 1987 Jan;53(1):29-31. No abstract available. PMID 3545399
- [Result] Tofoli GR, Ramacciato JC, de Oliveira PC, Volpato MC, Groppo FC, Ranali J. Comparison of effectiveness of 4% articaine associated with 1: 100,000 or 1: 200,000 epinephrine in inferior alveolar nerve block. Anesth Prog. 2003;50(4):164-8. PMID 14959904
- [Result] Sierra Rebolledo A, Delgado Molina E, Berini Aytis L, Gay Escoda C. Comparative study of the anesthetic efficacy of 4% articaine versus 2% lidocaine in inferior alveolar nerve block during surgical extraction of impacted lower third molars. Med Oral Patol Oral Cir Bucal. 2007 Mar 1;12(2):E139-44. PMID 17322803
- [Result] Wright GZ, Weinberger SJ, Marti R, Plotzke O. The effectiveness of infiltration anesthesia in the mandibular primary molar region. Pediatr Dent. 1991 Sep-Oct;13(5):278-83. PMID 1815200
- [Result] Ramadurai N, Gurunathan D, Samuel AV, Subramanian E, Rodrigues SJL. Effectiveness of 2% Articaine as an anesthetic agent in children: randomized controlled trial. Clin Oral Investig. 2019 Sep;23(9):3543-3550. doi: 10.1007/s00784-018-2775-5. Epub 2018 Dec 14. PMID 30552590

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04465149/Prot_SAP_000.pdf